CLINICAL TRIAL: NCT01775150
Title: Using Mobile Phone Text Messaging to Reduce Maternal and Infant Deaths in Remote Rural Areas in China
Brief Title: Saving Mother and Baby With Text Messaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian International Development Agency (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0029-01-04-01-01
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Bleeding; Infection; Malnutrition; Complications
Keywords: mobile phone text messaging; maternality; infant; death rate
MeSH Terms: conditions — Hemorrhage; Infections; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- health education (Experimental): health education via text messaging
  Interventions: Other: health education
- no health education (No Intervention): no health education via text messaging

INTERVENTIONS:
Other: health education — Health education via text messaging
  Arms: health education

SUMMARY:
We plan to integrate WHO educational material using mobile phone text messaging, target on pregnant women in remote rural areas in China. We hypothsized that text messaging can have major impact on reducing maternal and infant deaths in rural China because text messaging is accessible, acceptable, and affordable.

DETAILED DESCRIPTION:
1. Sampling method:

   Random sampling method will be used. Counties in Huaihua area of Chinese province of Hunan will be randomly allocated to intervention and non-intervention groups.
2. The intervention:

   Mobile phone text messages containing maternal and newborn health care education material will be sent to mothers-to-be at the first, second and third trimester, and again postpartum period.
3. Statistical analysis:

We will first compare the baseline characteristics (including the average income, adult educational level, and maternal and perinatal mortality rates in the past two years) between the 2 arms of experiment. For costs data, total costs, costs per participating woman, and costs per maternal/infant death avoided will be reported. For primary outcomes, we will determine and report rate ratios, risk differences, and numbers needed to treat (NNT) from the experimental arm (i.e., mobile phone text messaging), using the usual care arm (no text messaging) as the reference. Relative risks and 95% confidence intervals will be expressed as the effect measures. We will estimate the adjusted relative risks and 95% confidence intervals by regression analysis. Mixed models taking consideration of multi-level measures (e.g., mortality and morbidity measured at individual level and intervention measured at village level) will be used in the regression analysis (Donner and Klar, 2000).

ELIGIBILITY:
Inclusion Criteria:

* women who were registered by local Maternal Child Health unit during the study period

Exclusion Criteria:

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5646 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Neonatal death | 28 days
  28 days after birth

SECONDARY OUTCOMES:
Maternal death | 300 days
  From conception to 42 days postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Rihua Xie, PhD, Principal Investigator — Ottawa Hospital Research Institute; Shi Wu Wen, PhD, Study Director — Ottawa Hospital Resarch Institute
Locations (1):
- Ottawa Hospital Research Institue, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Xie RH, Tan H, Taljaard M, Liao Y, Krewski D, Du Q, Wen SW. The Impact of a Maternal Education Program Through Text Messaging in Rural China: Cluster Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Dec 19;6(12):e11213. doi: 10.2196/11213. PMID 30567693